CLINICAL TRIAL: NCT06477172
Title: A Multi-site, Prospective, Observational Study of Autologous Hair Follicle Secretome (aHFS) as an Adjunct to Medical Aesthetic Procedures
Brief Title: Autologous Hair Follicle Derived Secretome as Adjunct to Aesthetic Procedures
Status: Recruiting | Type: Observational
Sponsor: Acorn Biolabs Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ACN-101
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Post Procedural Erythema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-interventional, multi-site, prospective, open-label, observational, real-world study of autologous hair follicle secretome use.

DETAILED DESCRIPTION:
This non-interventional, observation study is to collect real-world data on the use of an autologous, hair follicle derived secretome topical cosmetic product following various medical aesthetic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* Ages: 18-60
* Any Fitzpatrick skin type
* Planning a medical aesthetic procedure
* For subjects receiving hair procedures:

  1. Androgenic alopecia
  2. Traction alopecia
  3. Scarring alopecia
  4. Stable use of any medication or supplement for hair loss, including finasteride, any other 5 α-reductase inhibitor, minoxidil, steroids, or hormonal products, during the 3 months prior to enrollment in the study is allowed.
  5. No intention to start new hair growth medications or change dose of hair growth medications from the time of consent through the end of the study follow-up period.
* Undergoing one of the following medical aesthetic procedures:

  1. Laser resurfacing of the face (ablative or non-ablative) or Ellacor of the face
  2. Microneedling of the face (roller, stamper, radiofrequency or pen) or Tixel of the face
  3. Microneedling of the scalp (roller, stamper or pen for hair loss) or Keralase of the scalp
  4. Surgery scars, either old or new as long as old scars are also being treated with ablative or non-ablative laser or microneedling (e.g. abdominoplasty, breast reduction/ reconstruction/enhancement, post-weight loss, etc.
* Planning to use Acorn Autologous Hair Follicle Secretome cosmetic product

Exclusion Criteria:

* Pregnant or Breastfeeding
* Participation in an interventional clinical trial in the last 30 days
* Use of other topical cosmetic products that may confound results
* Use of retinoids within 7 days prior to facial procedure
* For those receiving hair treatment, must not have had a hair transplant in the treatment area within the past 12 months
* Any health condition that in the investigator's opinion should preclude participation in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be patients planning a medical aesthetic procedure and use of Autologous Hair Follicle Secretome cosmetic post-procedure.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Post-Procedure Symptoms | 1-7 days
  Symptoms of redness, swelling, oozing, pain, tenderness, crusting, itching and discoloration will be measured using a 1-10 likert scale with 0 being best possible and 10 being worst imaginable.
Downtime Questionnaire | 1-7 days
  Questionnaire asking what activities would they have done, if it were not for their face appearance. Date of end of downtime captured.

CONTACTS AND LOCATIONS:
Overall Officials: Drew Taylor, PhD, Study Chair — Acorn Biolabs
Locations (29):
- United States (22):
  - BelleSante, Scottsdale, Arizona
  - Behr Laser & Skin Care Center, Fresno, California
  - Aesthetics By Dr. Lee, Granite Bay, California
  - Carlo Honrado, MD, FACS, Los Angeles, California
  - N2 Aesthetics, Manhattan Beach, California
  - Marina Plastic Surgery, Marina del Rey, California
  - M Beauty by Tess, San Diego, California
  - Dr. Christie, West Hollywood, California
  - Ziering Medical, West Hollywood, California
  - Bauman Medical, Boca Raton, Florida
  - Mirror Plastic Surgery, St. Petersburg, Florida
  - Hive Aesthetic LLC, Chicago, Illinois
  - Chernoff Cosmetic Surgery, Indianapolis, Indiana
  - AIEREM Aesthetics Spa & Plastic Surgery, Manhattan, New York
  - Lewis Dermatology and Associates, New York, New York
  - Unger Medical Hair Transplant Clinic, New York, New York
  - Sadick Dermatology, New York, New York
  - AIEREM Aesthetics Spa & Plastic Surgery, Syosset, New York
  - Austin Plastic Surgeon, Austin, Texas
  - Dallas Plastic Surgery Institute, Dallas, Texas
  - US Dermatology Partners / Dermatology Associates of Tyler, Tyler, Texas
  - AG Aesthetic Centre, Vancouver, Washington
- Canada (7):
  - Dr. Jean Carruthers Cosmedic, Vancouver, British Columbia
  - Dr. Amber Bocknek, Aurora, Ontario
  - Compass Dermatology, Toronto, Ontario
  - Rejuuv, Toronto, Ontario
  - Dr. Nowell Solish Cosmetic Dermatologist, Toronto, Ontario
  - BeSpoke Wellness, Toronto, Ontario
  - Clinique Antiaging, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No